CLINICAL TRIAL: NCT01121185
Title: A Phase II Randomized, Double-Blind, Placebo Controlled Study of the Clinical Effectiveness of a Human Monoclonal Antibody Against Hepatitis C Virus E2 Glycoprotein (MBL-HCV1) in Hepatitis C Infected Patients Undergoing Liver Transplantation
Brief Title: Study in Hepatitis C Virus (HCV) Infected Patients Undergoing Liver Transplantation to Evaluate a Human Monoclonal Antibody Against Hepatitis C
Acronym: MBL-HCV1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to slower than anticipated subject accrual.
Sponsor: MassBiologics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MBL-HCV1-10-02
Record Dates: First submitted 2010-05-06; First posted 2010-05-12 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-03

CONDITIONS: HCV Infection; Liver Transplantation
Keywords: Hepatitis C virus (HCV); Liver transplantation; Human Monoclonal Antibody
MeSH Terms: conditions — Hepatitis C | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBL-HCV1 (Experimental)
  Interventions: Biological: MBL-HCV1
- 0.9% sodium chloride (Placebo Comparator)
  Interventions: Other: 0.9% Sodium chloride Placebo

INTERVENTIONS:
Biological: MBL-HCV1 — 50 mg/kg MBL-HCV1, intravenous
  Arms: MBL-HCV1
Other: 0.9% Sodium chloride Placebo — 0.9% sodium chloride, intravenous
  Other Names: Normal Saline
  Arms: 0.9% sodium chloride

SUMMARY:
The purpose of this study is to determine whether a human monoclonal antibody against Hepatitis C (MBL-HCV1) is effective in preventing detectable levels of Hepatitis C virus in patients undergoing liver transplantation due to chronic HCV infection. The study will also determine if MBL-HCV1 is effective in delaying or reducing the amount of detectable HCV in patients after transplant.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo controlled study in Hepatitis C (HCV) infected patients undergoing liver transplantation. Chronically infected patients with HCV genotype 1a scheduled to receive a liver transplant from either a deceased or living donor who satisfy all study inclusion or exclusion criteria will be approached to participate. The study will be conducted in two parts to test a human monoclonal antibody against Hepatitis C (MBL-HCV1). In Part 1, sixteen eligible patients will be randomized 1:1 to receive 50 mg/kg MBL-HCV1 or 0.9% sodium chloride placebo intravenously. Eleven doses will be given during the first 14 days post transplantation. Patients will be evaluated through day 56 for safety and clinical outcomes that include measurement of anti-HCV antibodies, anti-drug antibody and HCV viral load. On study visit day 42, a liver biopsy will be performed for evaluation of hepatitis. Physical examination, vital sign measurements, emergence of adverse events and concomitant medication usage will be assessed at scheduled visits and as needed during the 56 day study period.

The Data Safety and Monitoring Board will perform a futility analysis after the first 16 patients have been enrolled and completed study follow-up through study visit day 42 post transplant. Based on the results of the interim analysis, the dose of MBL-HCV1 for part 2 of the study will be determined. Part 2 of the study will be conducted in the same manner as Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age with documented chronic hepatitis C virus infection of genotype 1a undergoing liver transplantation from either a deceased donor or living donor.
* Patient or legal guardian/health care proxy must have read, understood and provided written informed consent and HIPAA authorization after the nature of the study has been fully explained.

Exclusion Criteria:

* Positive serology for Hepatitis B surface Antigen
* Positive serology for HIV
* Pregnancy or breastfeeding
* Previous history of any organ transplant
* Planned receipt of combined organ transplant (e.g. liver and kidney)
* Receipt or planned receipt of immune globulin (IVIG) within 90 days of enrollment
* History of extrahepatic malignancy and/or receiving chemotherapy within 90 days prior to enrollment with the exception of chemoembolization for hepatocellular carcinoma
* Hepatocellular carcinoma with tumor burden outside of the Milan criteria
* History of chronic renal insufficiency or creatinine > 2.5 for ≥ six months
* Personal or family history of deep venous thrombosis or pulmonary embolism
* Receipt of liver allograft from HCV positive donor or Hepatitis B core antibody positive donor
* Receipt of liver allograft donated after cardiac death of donor
* Receipt of any antiviral agents, licensed or investigational for hepatitis C virus within 90 days prior to enrollment
* Receipt of any other investigational study product within 30 days prior to enrollment
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the patient participating in the study or make it unlikely that the patient could complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah C. Molrine, MD, Study Director — Massbiologics of University of Massachusetts Medical School
Locations (8):
- United States (8):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Methodist Healthcare Foundation, Memphis, Tennessee

REFERENCES:
- [Result] Chung RT, Gordon FD, Curry MP, Schiano TD, Emre S, Corey K, Markmann JF, Hertl M, Pomposelli JJ, Pomfret EA, Florman S, Schilsky M, Broering TJ, Finberg RW, Szabo G, Zamore PD, Khettry U, Babcock GJ, Ambrosino DM, Leav B, Leney M, Smith HL, Molrine DC. Human monoclonal antibody MBL-HCV1 delays HCV viral rebound following liver transplantation: a randomized controlled study. Am J Transplant. 2013 Apr;13(4):1047-1054. doi: 10.1111/ajt.12083. Epub 2013 Jan 28. PMID 23356386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with HCV genotype 1a infection scheduled to undergo liver transplantation were recruited at 8 U.S. transplantation centers between June 2010 and April 2011. Due to slower than anticipated subject accrual, enrollment was stopped after 13 subjects were randomized; 11 underwent liver transplantation and received the study intervention.
Pre-assignment Details: Reasons for exclusion after randomization included identification of a protocol-specified exclusion criterion in the recipient or the donor at the time of organ offer or failure to undergo liver transplantation.
Groups:
- Experimental: MBL-HCV1: Eleven intravenous infusions of MBL-HCV1 (50 mg/kg) human monoclonal antibody administered during the first 14 days post-transplantation: three infusions were given on Day 0 (1-4 hours prior to anhepatic phase, during the anhepatic phase, and within 4-12 hours post-reperfusion), daily infusions were administered on days 1 through 7, and the final infusion was given on day 14 ± 2 post transplantation.
- Placebo Comparator: 0.9% Sodium Chloride: Eleven intravenous infusions of 0.9% sodium chloride administered during the first 14 days post-transplantation: three infusions were given on Day 0 (1-4 hours prior to anhepatic phase, during the anhepatic phase, and within 4-12 hours post-reperfusion), daily infusions were administered on days 1 through 7, and the final infusion was given on day 14 ± 2 post transplantation.
Period: Overall Study
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Started | 7 | 6
Infused | 7 | 5 (Excluded medical condition identified in one subject after randomization but before study infusion.)
Transplanted | 6 (One subject initiated the first study infusion, but transplant surgery was subsequently cancelled.) | 5
Completed | 6 | 5
Not Completed | 1 | 1
Not completed — Not infused | 0 | 1
Not completed — Not transplanted | 1 | 0

BASELINE CHARACTERISTICS:
Population: The eleven subjects who were randomized, initiated study infusions, and underwent liver transplantation were included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 60.9 [55.9 to 66.6] | 57.2 [53.5 to 60.3] | 59.2 [53.5 to 66.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Hepatocellular carcinoma [Number; unit: participants] | 4 | 2 | 6
Serum HCV RNA concentration [Median (Full Range); unit: log10 IU/mL] | 6.07 [4.47 to 7.19] | 5.59 [5.12 to 6.58] | 6.03 [4.47 to 7.19]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Detectable Serum HCV RNA at Day 42 Post-Transplantation
Description: Serum HCV RNA was measured by Quantitative RT-PCR
Time Frame: At Day 42 post-transplantation
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
percentage of participants | 100 | 100

2. Secondary Outcome: The Incidence of Adverse Events and Treatment-Emergent Adverse Events Determined Through Medical History, Physical Examination and Laboratory Evaluation
Description: Adverse events were assessed by targeted medical history, physical examinations and laboratory testing. Subjects were asked at scheduled study visits through day 42 whether they experienced solicited adverse reactions (fever, chills, nausea, rash, joint pain or swelling, shortness of breath, headache, fatigue, and hives). In addition to these solicited adverse events, subjects were asked at all scheduled study visits through day 56 to report any other adverse events, regardless of whether the event was thought to be related to the study infusions. Adverse events were summarized by System Organ Class (SOC) using MedDRA (version 12.0)
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Number; unit: events
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
events
  General Disorders And Administration Site Conditio | 13 | 6
  Gastrointestinal Disorders | 9 | 9
  Metabolism And Nutrition Disorders | 7 | 10
  Investigations | 16 | 7
  Nervous System Disorders | 7 | 3
  Skin And Subcutaneous Tissue Disorders | 3 | 4
  Injury, Poisoning And Procedural Complications | 4 | 3
  Respiratory, Thoracic And Mediastinal Disorders | 3 | 2
  Renal And Urinary Disorders | 4 | 1
  Psychiatric Disorders | 3 | 1
  Vascular Disorders | 2 | 1
  Blood And Lymphatic System Disorders | 1 | 2
  Infections And Infestations | 1 | 9
  Eye Disorders | 1 | 1
  Musculoskeletal And Connective Tissue Disorders | 2 | 1
  Hepatobiliary Disorders | 1 | 0
  Reproductive System And Breast Disorders | 1 | 0
  Ear And Labyrinth Disorders | 0 | 1

3. Secondary Outcome: Change in Serum HCV RNA Between Baseline and Day 3, 14, 28 and 42 Post-Transplantation
Description: Serum HCV RNA was measured by quantitative RT-PCR. The change in HCV RNA from baseline was obtained by calculating the difference between the baseline pre-transplantation HCV RNA level and the HCV RNA level measured at each study visit.
Time Frame: Baseline and Day 3, 14, 28 and 42 Post-Transplantation
Population: as for baseline characteristics
Measure: Median (Full Range); unit: log10 IU/mL
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
log10 IU/mL
  Day 3 | -3.07 [-3.45 to -2.17] | -1.01 [-2.87 to 1.03]
  Day 14 | -2.48 [-3.77 to 0.81] | 0.10 [-2.60 to 2.09]
  Day 28 | -0.75 [-3.23 to 1.01] | 1.22 [-2.00 to 2.59]
  Day 42 | 0.23 [-1.16 to 0.93] | 1.22 [-2.14 to 2.72]

4. Secondary Outcome: Histologic Evidence of Hepatitis by Histologic Activity Index (HAI) Score at Baseline and Day 42
Description: Liver biopsies obtained at baseline (day 0) and day 42 post-transplantation were assessed for histologic evidence of hepatitis by a pathologist blinded to treatment assignment using the Ishak modification of the Knodell histologic grading system to assign a histologic activity index (HAI) score. The HAI score consists of a sum of four components: 1) periportal or periseptal interface hepatitis; 2) confluent necrosis; 3) focal lytic necrosis, apoptosis and focal inflammation; 4) portal inflammation. The total HAI score can range from a minimum of 0 to a maximum of 18, with higher scores indicating more severe hepatic inflammation.
Time Frame: Baseline Day 0 and Day 42
Population: The 11 subjects who were randomized, initiated study infusions, and underwent transplantation were included in the analysis population. On day 0, all subjects had pre-transplant biopsy specimens available for analysis. On day 42, 4 subjects in the MBL-HCV1 group and 5 subjects in the placebo group had biopsy specimens available for analysis.
Measure: Median (Full Range); unit: Histologic activity index (HAI) score
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
Histologic activity index (HAI) score
  Day 0 | 0.0 [0 to 0] | 1.0 [0 to 2]
  Day 42 | 0.6 [0 to 1] | 4.0 [1 to 6]

5. Secondary Outcome: Graft Function Assessed by Measurement of Biochemical and Synthetic Function at Multiple Time Points / International Normalized Ratio (INR)
Description: Biochemical function was assessed by measurement of alanine aminotransferase (ALT) and total bilirubin and synthetic function was assessment by measurement of the pro-thrombin time (reported as the international normalized ratio, INR) at multiple time-points during the 56-day study period. The table below displays the INR at each time-point. The INR is the ratio of a patient's prothrombin time to a control sample, raised to the power of the ISI value (International Sensitivity Index) for the batch of tissue factor being used for the assay.
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: unitless
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
unitless
  Screening | 1.5 [1 to 2.3] | 1.5 [0.97 to 2.9]
  Day 0 | 1.6 [1.1 to 2.7] | 1.5 [1 to 2.9]
  Day 1 | 1.4 [1.1 to 1.6] | 1.3 [1.1 to 1.6]
  Day 2 | 1.2 [1 to 1.4] | 1.3 [1 to 1.6]
  Day 3 | 1.2 [0.9 to 1.6] | 1.1 [1 to 1.2]
  Day 4 | 1.5 [0.9 to 3.3] | 1.1 [1 to 1.2]
  Day 5 | 1.6 [0.9 to 4] | 1.1 [1.1 to 1.2]
  Day 6 | 1.4 [0.9 to 2.7] | 1.2 [1.05 to 1.2]
  Day 7 | 1.3 [1 to 2.2] | 1.1 [0.99 to 1.3]
  Day 14 | 1.2 [1 to 1.7] | 1.1 [0.95 to 1.2]
  Day 21 | 2 [1.1 to 3.7] | 1.1 [0.96 to 1.2]
  Day 28 | 1.6 [1 to 3] | 1.1 [0.93 to 1.2]
  Day 42 | 1.2 [1 to 1.6] | 1.1 [0.98 to 1.2]
  Day 56 | 1.1 [1 to 1.2] | 1.1 [1 to 1.3]

6. Secondary Outcome: Graft Function Assessed by Measurement of Biochemical and Synthetic Function at Multiple Time Points / Alanine Aminotransferase (ALT)
Description: Biochemical function was assessed by measurement of alanine aminotransferase (ALT) and total bilirubin and synthetic function was assessment by measurement of the pro-thrombin time (reported as the international normalized ratio, INR) at multiple time-points during the 56-day study period. The table below displays the ALT at each time-point.
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: U/L
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
U/L
  Screening | 74 [46 to 107] | 114 [60 to 263]
  Day 0 | 76 [44 to 111] | 107 [71 to 164]
  Day 1 | 565 [90 to 1571] | 404 [88 to 832]
  Day 2 | 501 [75 to 1084] | 415 [87 to 986]
  Day 3 | 374 [62 to 799] | 464 [80 to 1385]
  Day 4 | 301 [56 to 572] | 355 [57 to 975]
  Day 5 | 243 [57 to 421] | 253 [49 to 626]
  Day 6 | 207 [50 to 295] | 219 [43 to 495]
  Day 7 | 163 [48 to 208] | 176 [37 to 338]
  Day 14 | 38 [15 to 77] | 54 [21 to 116]
  Day 21 | 34 [13 to 60] | 55 [15 to 141]
  Day 28 | 21 [7 to 26] | 109 [18 to 232]
  Day 42 | 22 [14 to 32] | 174 [14 to 426]
  Day 56 | 41 [23 to 96] | 183 [19 to 606]

7. Secondary Outcome: Graft Function Assessed by Measurement of Biochemical and Synthetic Function at Multiple Time Points / Total Bilirubin
Description: Biochemical function was assessed by measurement of alanine aminotransferase (ALT) and total bilirubin and synthetic function was assessment by measurement of the pro-thrombin time (reported as the international normalized ratio, INR) at multiple time-points during the 56-day study period. The table below displays the total bilirubin at each time-point.
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
mg/dL
  Screening | 2.8 [1.2 to 5] | 8.9 [0.57 to 33.7]
  Day 0 | 2.6 [0.8 to 4.1] | 2.9 [0.64 to 5.5]
  Day 1 | 3.3 [0.8 to 6.1] | 4.7 [2.07 to 10.1]
  Day 2 | 2.3 [1.1 to 3.1] | 4.1 [1.76 to 8.7]
  Day 3 | 2 [1.2 to 3.1] | 4.7 [1.72 to 9.1]
  Day 4 | 2 [1.4 to 2.8] | 5.5 [1.44 to 10.9]
  Day 5 | 2.1 [1.3 to 3.6] | 7 [1.47 to 12.5]
  Day 6 | 2.6 [1.3 to 5.1] | 8.3 [1.22 to 17.1]
  Day 7 | 3 [1 to 9.2] | 8.2 [1.11 to 19]
  Day 14 | 1.2 [0.7 to 2.7] | 2.6 [0.49 to 4.9]
  Day 21 | 1 [0.6 to 2] | 1.7 [0.37 to 2.8]
  Day 28 | 0.9 [0.5 to 1.4] | 1.5 [0.27 to 2.4]
  Day 42 | 0.8 [0.5 to 1.1] | 1.2 [0.29 to 1.9]
  Day 56 | 0.7 [0.4 to 0.9] | 2 [0.16 to 5.3]

8. Secondary Outcome: Time to Onset of Recurrence of Detectable HCV RNA Post-Transplantation
Description: Serum HCV RNA was measured by Quantitative RT-PCR
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Number; unit: days
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
days | NA — The planned analysis could not be performed because an insufficient number of participants had undetectable HCV RNA post-transplantation. A post-hoc analysis of time to virologic rebound (≥ 1 log10 increase above viral nadir) was performed. | NA — The planned analysis could not be performed because an insufficient number of participants had undetectable HCV RNA post-transplantation. A post-hoc analysis of time to virologic rebound (≥ 1 log10 increase above viral nadir) was performed.

9. Post Hoc Outcome: Time To Viral Rebound Post-Transplantation(Serum HCV RNA Increased ≥ 1 log10 From Viral Nadir)
Description: The time of viral rebound was defined as the time of the first measurement of serum HCV RNA increased ≥ 1 log10 from the viral nadir (the lowest serum HCV RNA level post-transplantation). Serum HCV RNA was measured by RT-PCR.
Time Frame: Through Day 56
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: days
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Number analyzed (Participants) | 6 | 5
days | 22.7 [15.0 to 34.4] | 2.33 [1.18 to 3.10]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the start of the first infusion through day 56 post-transplantation
Description: Adverse events were assessed by history, physical examinations and laboratory testing through day 56. In addition, the following adverse reactions were specifically solicited through day 42: fever, chills, nausea, rash, joint pain or swelling, shortness of breath, headache, fatigue, and hives.
Arm/Group | Experimental: MBL-HCV1 | Placebo Comparator: 0.9% Sodium Chloride
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: MBL-HCV1 (N=6) | Placebo Comparator: 0.9% Sodium Chloride (N=5)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 2 (2)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Blood Glucose Fluctuation (Investigations) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: MBL-HCV1 (N=6) | Placebo Comparator: 0.9% Sodium Chloride (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Generalised Oedema (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Norovirus (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Albumin Urine Present (Investigations) | 1 (1) | 0 (0)
Bacterial Test Positive (Investigations) | 0 (0) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0)
Blood Bilirubin Increased (Investigations) | 2 (2) | 0 (0)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0)
Blood Magnesium Decreased (Investigations) | 1 (1) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0)
Clostridium Difficile Toxin Test (Investigations) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 3 (3) | 2 (2)
Urinary Casts (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 2 (2)
Peroneal Nerve Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Reperfusion Injury (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less